CLINICAL TRIAL: NCT04879940
Title: Phase II Study to Evaluate the Safety and Efficacy of Prostatic Artery Embolization in Patients With Localized Prostate Carcinoma and Obstructive Lower Urinary Tract Symptoms
Brief Title: Phase II Study to Evaluate the Safety and Efficacy of Prostatic Artery Embolization
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-20832
Record Dates: First submitted 2021-05-05; First posted 2021-05-10 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Prostate Carcinoma; Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Hyperplasia | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Prostatic Artery Embolization (PAE) (Experimental): Participants who receive PAE with Merit Medical Embospheres.
  Interventions: Device: Merit Medical Embospheres; Radiation: Radiation Therapy

INTERVENTIONS:
Device: Merit Medical Embospheres — Prostatic Artery Embolization will performed as an outpatient procedure in Interventional Radiology. Bilateral selective pelvic angiograms will be performed to localize the prostatic arteries. Cone-beam or 3D computed tomography (CT) will be performed prior to embolization, if technically feasible and necessary. Embolization will be performed using Merit Medical Embospheres.
Radiation: Radiation Therapy — Patients will undergo standard of care definitive radiation therapy.

SUMMARY:
This is a Phase II prospective clinical trial in which patients with prostate carcinoma and obstructive lower urinary tract symptoms electing for radiation therapy will undergo Prostatic Artery Embolization (PAE) prior to treatment. PAE will be administered by Interventional Radiology. Patients will be seen for follow-up at 6 weeks and 12 weeks following PAE after which they will start definitive radiotherapy. After completion of radiotherapy the patient will be seen at 12 weeks

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed prostate adenocarcinoma in the very low or low or favorable intermediate risk risk stratification groups (i.e. Gleason Grade groups 1 and 2) who are eligible for and who select XRT as their cancer management method.
* Ability to receive prostatic artery embolization within 6-12 weeks of definitive radiation therapy.
* Ability to understand and the willingness to sign a written informed consent document
* Prostate larger than 60 grams but less than 150 grams, as assessed by imaging scans
* American Urologic Association (AUA) or International Prostate Symptom Score (IPSS) Score ≥ 15
* Normal organ and marrow function as defined in protocol

Exclusion Criteria:

* Patients with Gleason Grade Group 1 or 2 PCa who select active surveillance as their cancer management method.
* Receiving androgen deprivation therapy (ADT)
* Patients with unfavorable intermediate (Gleason Grade Group 3) or high risk localized PCa (Gleason Grade Groups 4 and 5)
* Receiving any investigational agents for the explicit purpose of prostatic size reduction
* Inability to receive prostatic artery embolization (PAE) within 6-12 weeks of definitive radiation therapy
* Active urinary tract infection (UTI)
* History of severe allergic reaction to intravenous contrast media (iodinated and gadolinium- based) or any agents used during the PAE; patient cannot be medicated against allergic reaction prior to PAE.
* Active cystolithiasis or prostatitis
* Inability to have multi-parametric magnetic resonance imaging (mpMRI)
* Prior transurethral resection of the prostate (TURP) within 2 years
* Prostate size greater than or equal to150 grams
* Vulnerable subjects (e.g., inmates and developmentally delayed adults) who are subjects for whom the study may be unsafe or whose rights may be violated with enrollment.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male
Enrollment: 26 (Estimated)
Dates: Start 2022-02-23 (Actual); Primary Completion 2026-01-01 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in International Prostate Symptom Score | At screening, Day of PAE, and 6 weeks & 12 weeks after PAE
  Participants will take quality of life questionnaires including the International Prostate Symptom Score (IPSS)questionnaire to determine changes in prostate symptoms. Questionnaire will be taken at screening, Day 0- day of prostatic artery embolization (PAE), and at 6 weeks and 12 weeks after PAE. The IPSS asks the patient to rate urinary symptoms on a scale of 0-5, 0 indicating the participant has not had a symptom at all, and 5 indicating the symptom "almost always".

SECONDARY OUTCOMES:
Prostate Volume Reduction after PAE | At 12 weeks
  Prostate volume will be determined by MRI prior to PAE and at 12 weeks post PAE to determine changes in volume.
Change in American Urologic Association Score | At 18 weeks
  Participants will take quality of life questionnaires including the American Urologic Association (AUA) test to assess genitourinary toxicity after PAE and radiation therapy. The AUA questionnaire asks the patient to rate urinary symptoms on a scale of 0-5, 0 indicating indicating the participant has not had a symptom at all, and 5 indicating the symptom "almost always".

CONTACTS AND LOCATIONS:
Overall Officials: Nainesh S Parikh, MD, MBA, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No